CLINICAL TRIAL: NCT00475358
Title: Efficacy and Safety of Duloxetine Compared With Placebo in Subjects With Stress Urinary Incontinence
Brief Title: Efficacy and Safety Stress Urinary Incontinence Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6231; F1J-MC-SBBT
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine
Drug: Placebo

SUMMARY:
Study F1J-MC-SBBT will examine the effect of duloxetine treatment in women with SUI. The inclusion and exclusion criteria of this Phase 3 study will ensure that all subjects have a clinical diagnosis of SUI.

ELIGIBILITY:
Inclusion Criteria:

* Are greater than 20 years of age.
* Are female outpatients.
* Present with SUI based on the disease diagnostic criteria, average at least one incontinent episode per day on the screening diary, and have had symptoms of SUI for a minimum of 3 months prior to study entry.
* Are women of non-childbearing potential by reason of hysterectomy, other surgery, or natural menopause, or are women of childbearing potential who test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a medically accepted means of contraception (for example, intrauterine device [IUD], oral or injectable contraceptives, implant, barrier device, sterilization, abstinence, or sex with a vasectomized male partner) for the duration of the study. Women using oral contraceptives or hormone replacement therapy must have a stable dose and regimen for greater than or equal to 3 months prior to entry into the study.
* Have no language barrier, agree to comply with the requirements of the protocol, and sign a written informed consent document prior to entry into the study.

Exclusion Criteria:

* Suffer from severe constipation (for example, have impacted rectum at time of physical examination despite recent evacuation).
* Has a physical examination, neurological and/or vaginal examination results which, in the opinion of the investigator, should exclude the subject.
* Are on a medication regimen (including diuretics) for which dose and/or frequency has not been stable for at least 12 weeks prior to randomization, or is anticipated to change during the course of the study.
* Have had any major inpatient surgery within 3 months prior to study entry.
* Have current diagnosis of any of the following conditions, disorders, or diseases of the genito-urinary tract: Ureteric, bladder, urethral, or rectal fistula
* Uncorrected congenital abnormality leading to urinary incontinence
* Detrusor instability or noncompliant bladder
* Adult enuresis
* Voiding difficulty (i.e., subject complains of difficulty emptying their bladder).

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-04; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
To assess efficacy of duloxetine 80 mg/day for 8 weeks in women with stress urinary incontinence (SUI) compared with placebo as measured by percent change in incontinence episode frequency from baseline.

SECONDARY OUTCOMES:
To compare the efficacy of duloxetine with that of placebo as measured by the change in the disease-specific quality of life instrument (I QOL) scores from baseline to endpoint.
To compare the efficacy of duloxetine with that of placebo in subject perceived improvement in SUI as measured by the Patient's Global Impressions of Improvement (PGI I) questionnaire.
To compare the safety of duloxetine with that of placebo in the treatment of SUI based on vital signs, laboratory values, and the occurrence of treatment-emergent adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District, Taiwan

REFERENCES:
- [Derived] Lin AT, Sun MJ, Tai HL, Chuang YC, Huang ST, Wang N, Zhao YD, Beyrer J, Wulster-Radcliffe M, Levine L, Chang C, Viktrup L. Duloxetine versus placebo for the treatment of women with stress predominant urinary incontinence in Taiwan: a double-blind, randomized, placebo-controlled trial. BMC Urol. 2008 Jan 25;8:2. doi: 10.1186/1471-2490-8-2. PMID 18221532
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com